CLINICAL TRIAL: NCT05309577
Title: Self-Care for Dementia Caregivers Using the myRhythmWatch
Brief Title: Self-Care for Dementia Caregivers
Acronym: Care2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Activity Rhythm Solutions Corporation (Unknown); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sarah T. Stahl, PhD, Associate Professor of Psychiatry and Clinical and Assistant Professor of Translational Science, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY21060122; P30AG024978 (NIH); R41AG069596 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Aging; Mental Disorder; Eating, Healthy; Physical Inactivity; Prodromal Symptoms; Sleep; Alzheimer Disease; Dementia; Circadian Rhythm Disorders
Keywords: Caregivers; Carers; Alzheimer Disease; Alzheimer Dementia; Dementia; Twenty-Four Hour Rhythm; Geriatrics; Self Care; Circadian Rhythm
MeSH Terms: conditions — Mental Disorders; Sedentary Behavior; Prodromal Symptoms; Alzheimer Disease; Dementia; Chronobiology Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver Intervention (Experimental): Behavioral self-monitoring of sleep and activity up to 6 weeks, using the myRhythmWatch app, and motivational health coaching.
  Interventions: Behavioral: Behavioral Self-Monitoring + Motivational Interviewing

INTERVENTIONS:
Behavioral: Behavioral Self-Monitoring + Motivational Interviewing — Participants (n=20) will wear a iWatch to continuously measure their objective sleep-wake activity. The iWatch data sync to the new myRhythmWatch app, where participants will monitor their behavioral rhythm. Participants will also interact with a 'health coach' about their recorded behaviors weekly. This health coach will use motivational interviewing to enhance older adult caregivers' confidence and intrinsic motivation to engage in regular self-care.

SUMMARY:
The Self-care for Dementia Caregivers Study is a behavioral health intervention that uses digital monitoring tools and motivational health coaching to help caregivers of persons with dementia engage in a regular routine of sleep and activity. Participants wear an apple watch for the objective collection of sleep-wake rhythms. They receive personalized feedback on their sleep-wake rhythms via a new app. Health coaches call participants weekly, for up to 6 weeks to help participants meet their health/sleep goals and promote self-knowledge of regular routines. Participants will help the study team improve the design elements and content of the mobile app. The goal of this intervention is to reduce depressive and insomnia symptoms.

DETAILED DESCRIPTION:
Caregivers of family members with Alzheimer's Disease (AD) and AD-related dementias (ADRD) experience high rates of psychological stress, physical impairments, and often, disruptions in normal daily activities. Caregivers must be alert both at night and during the day, and often on an inconsistent schedule. As a result, caregivers are less likely to sleep, exercise, and be socially active on a regular schedule. Disruptions of these biological and behavioral time cues, or "zeitgebers", in turn decrease the stability of the body's biological clock, placing caregivers at high risk for adverse health outcomes related to an out-of-sync biological clock (e.g. diabetes, cardiovascular disease, and depression, among others). Caregivers of individuals with ADRD experience worse health outcomes compared with other types of caregivers, likely due to more heavily or frequently disrupted schedules.

For this research study, up to 25 individuals aged 50 and older who are providing care for a family member with mild-to-moderate dementia will be included. Data from 5 participants will be used for the development of an intervention manual (NIH Stage Model IA). A small pilot study will be conducted (NIH Stage Model IB) in which 20 participants will use a new mobile app - my rhythm watch - for up to 6 weeks. Objective actigraphic measures of the 24-hour pattern of sleep and daytime activity - known as the circadian rest-activity rhythm (RAR) - will be measured continuously via the apple watch to evaluate circadian rhythms as a potential intervention target/mechanism of action. The investigators will measure the regularity, timing, and amplitude of behavioral patterns over a 24-hour period. Participants will be assessed at baseline, post-intervention, and 3-months post-intervention. Initially our plan was to focus an intervention on promoting self-care and reducing caregiving burden. However, in designing the trial, we switched the focus to the circadian-informed, behavioral activation-based approach that aimed to improve sleep and mood in caregivers. Therefore, the two main outcomes of interest were measures of depression symptom severity and insomnia symptom severity.

The study as described in the original registration (April 2022) never proceeded. The registration has been revised to reflect the study as modified after securing a technology partner (per funding requirements) and prior to study initiation

ELIGIBILITY:
Inclusion criteria for ADRD patients include:

* being ≥60 years
* having been diagnosed with Alzheimer's disease, vascular dementia, mixed Alzheimer's/vascular dementia, or frontotemporal dementia
* living with their caregiver
* being willing to wear the watch and participate in assessments and calls

Inclusion criteria for ADRD caregivers include:

* being a primary caregiver for an ADRD patient
* being ≥50 years
* experiencing stress/strain related to caregiving
* the person being cared for has problems with sleep or keeping a consistent routine
* scoring ≥5 on the PHQ-9 (experiencing depression symptoms)
* living with their care recipient
* being willing to try the app and participate in assessments and calls

Exclusion criteria for ADRD patients include:

* being less than 60 years
* not having a diagnosis of ADRD
* not living with their caregiver
* not being willing to wear the watch and participate in assessments and calls

Exclusion criteria for ADRD caregivers include:

* being less than 50 years
* not experiencing stress/strain related to caregiving
* the person being cared for does not have problems with sleep or keeping a consistent routine
* scoring <5 on the PHQ-9
* not living with their care recipient
* not being willing to try the app and participate in assessments and calls

Participants of this study may enroll as care givers or recipient-caregiver dyads.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah T Stahl, PhD, Principal Investigator — University of Pittsburgh, Assistant Professor of Psychiatry and Clinical and Translational Science
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be available, after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: De-identified individual participant date will be available indefinitely following publication. It may be shared with researchers who provide a methodologically sound proposal for the purpose of achieving the aims in the approved proposal. Proposals should be directed to sts80@pitt.edu. Approved requestors will need to sign a data access management agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited dementia caregivers (CG) from university-affiliated research registries. Eligible/interested dementia caregivers were screened for whether their care recipients, a person with dementia (PWD), would be eligible/interested in using the myRW app to track and monitor daily rhythms. Of the 25 dementia CGs we screened, 15 CGs were enrolled and allocated to the intervention; and 6 PWD were included in the intervention rendering a total sample of 21.
Pre-assignment Details: This single-arm pilot trial enrolled participants between March 2023 and April 2024 in Pittsburgh, PA.
Groups:
- Behavioral Intervention (Caregivers): Rest-activity rhythm monitoring via the myRW app plus motivational interviewing techniques to optimize rhythms in older dementia caregivers.
- Behavioral Intervention (PWD): Rest-activity rhythm monitoring via the myRW app to optimize rhythms in older persons with dementia (PWD).
Period: Overall Study
Arm/Group | Behavioral Intervention (Caregivers) | Behavioral Intervention (PWD)
Started | 15 | 6
Completed | 15 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Health outcomes were based on data from 15 dementia caregivers
Groups:
- Behavioral Intervention (PWD): Rest-activity rhythm monitoring via the myRW app plus motivational interviewing techniques to optimize rhythms in persons with dementia (PWD).
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention (Caregivers) | Behavioral Intervention (PWD) | Total
Number analyzed (Participants) | 15 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years
  years | 61.78 (8.40) | 81.45 (8.46) | 66.62 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants] — Participant sex
  Participants
    Female | 13 | 4 | 17
    Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 1 | 5
    White | 9 | 5 | 14
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported Ethnicity
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 15 | 6 | 21
    Unknown or Not Reported | 0 | 0 | 0
Depression symptoms [Mean (Standard Deviation); unit: score on a scale] — Depressive score on the Patient Health Questionnaire-9
  score on a scale | 6.64 (5.00) | 6.80 (7.40) | 6.68 (5.50)
Insomnia symptoms [Mean (Standard Deviation); unit: score on a scale] — Insomnia score on the Insomnia Severity Index
  score on a scale | 11.43 (5.10) | 8.60 (5.41) | 10.68 (5.19)

OUTCOME MEASURES:

1. Primary Outcome: Pre/Post Change in Depressive Symptoms
Description: The 9-item Patient Health Questionnaire (PHQ-9) scale is a self-reported questionnaire to be completed by the participant that assesses severity of depression. The PHQ-9 will be administered throughout the study to assess changes in depressive symptoms pre- and post-intervention. A minimum score on this metric is a 0, indicating no impact to patient health, and ranges up to a maximum score of 27, indicating more severe impacts to patient health.
Time Frame: Up to 6 weeks
Population: Eleven of the 15 caregivers completed pre-and post-treatment assessments and were included in the health outcome analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Behavioral Intervention: Rest-activity rhythm monitoring via the myRW app plus motivational interviewing techniques to optimize rhythms.
Arm/Group | Behavioral Intervention
Number analyzed (Participants) | 11
score on a scale | 2.27 (2.61)

2. Primary Outcome: Pre/Post Change in Insomnia Symptoms
Description: The 7-item Insomnia Severity Index (ISI) is a self-reported questionnaire to be completed by the participant that assesses severity of insomnia. The ISI will be administered throughout the study to assess changes in insomnia symptoms pre- and post-intervention. A minimum score on this metric is a 0, indicating no impact to patient health, and ranges up to a maximum score of 28, indicating more severe impacts to patient health.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention
Number analyzed (Participants) | 11
score on a scale | 5.64 (5.73)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 3 months
Description: We monitored all caregivers (n=15) for self-reported adverse events (AEs) using an AE reporting form. AEs were subsequently rated for severity and their relationship to study participation and coded using the NIH categorization of adverse events.
Groups:
- Behavioral Intervention (PWD): Rest-activity rhythm monitoring via the myRW app to optimize rhythms in persons with dementia (PWD).
Arm/Group | Behavioral Intervention (Caregivers) | Behavioral Intervention (PWD)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6
Other Adverse Events (participants affected / at risk) | 0/15 | 0/6

LIMITATIONS AND CAVEATS:
Due to cost restraints and the early phase nature of this study, we used a single-arm design. This precludes inference on the extent to which the observed health benefits were due to via real-time RAR monitoring, rather than other aspects of the intervention sessions, or non-specific therapeutic responses. Our sample consisted of adults willing/able to use digital technologies. Feasibility may be lower in adults with lower levels of technology literacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-11-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT05309577/Prot_001.pdf
  • Informed Consent Form (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT05309577/ICF_000.pdf